CLINICAL TRIAL: NCT01509911
Title: A Clinical Trial of Anti-Angiogenic Drug Combination Tl-118 for Pancreatic Cancer Patients Who Are Starting Gemcitabine Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tiltan Pharma Ltd. (Industry)
Collaborators: Technostat (Unknown); Novatrials (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLH-206
Record Dates: First submitted 2012-01-05; First posted 2012-01-13 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — TL-118; Gemcitabine

ARMS (2):
- TL-118 with standard of care Gemcitabine (Experimental)
  Interventions: Drug: TL-118
- Gemcitabine with out TL-118 (Active Comparator)
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: TL-118 — TL-118 investigational product is supplied as an oral liquid for daily administration at a specific dosing regimen. Treatment protocol includes weekly therapy cycles.
  Arms: TL-118 with standard of care Gemcitabine
Drug: Gemcitabine — Monthly cycles of 3 weekly treatments a month and one week off of treatment
  Other Names: Gemzar
  Arms: Gemcitabine with out TL-118

SUMMARY:
TL-118 is an anti-angiogenic drug combination designed for the treatment of cancer. The investigational product Tl-118 comprises of four well-known active components. The therapy is administrated at a unique dosing regimen that was found to be effective and advantageous in terms of safety. The product is formulated as an oral suspension, conveniently administrated by the patients at home and not requiring medical staff assistance. This Phase II clinical trial aims to evaluate the efficacy, safety and tolerability of TL-118 in Gemcitabine treated Pancreatic Cancer patients

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years at enrollment.
2. Metastatic Pancreatic Cancer
3. The patient has histologically or cytologically confirmed pancreatic adenocarcinoma.
4. Patient has measurable disease by (RECIST).
5. Patient is starting standard of care Gemcitabine treatment
6. ECOG performance status ≤ 1
7. Adequate renal function
8. Adequate hepatic function
9. Adequate bone marrow reserve
10. Resolution of prior therapy acute adverse events.
11. Patient is capable of swallowing.
12. Patient's Informed Consent. -

Exclusion Criteria:

1. Hypersensitivity to one or more of the TL-118 active components
2. Known Glucose-6-phosphate-dehydrogenase deficiency (G6PD).
3. CNS or Brain metastases
4. Prior systemic therapy for pancreas cancer
5. Subjects who received any investigational medication, prior local therapy for pancreas cancer , or any significant change in treatment within 1 month prior to screening
6. Concurrent use of any other investigational product
7. Subjects with a clinically significant or unstable medical condition that would preclude safe and complete study participation
8. Use of supplements or complementary medicines/botanicals, except for conventional multivitamin supplements, calcium, selenium and soy supplements.
9. Patient has known historical or active infection with HIV, hepatitis B, or hepatitis C
10. Circumstances likely to interfere with absorption of orally administrated drugs.
11. History of noncompliance to medical regimens or coexisting -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-01; Primary Completion 2016-10 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate as defined by Percentage of patients experiencing a Complete Response or a Partial Response or a Stable Disease according to RECIST measured at 16 weeks after treatment initiation | 16 weeks after treatment initiation

SECONDARY OUTCOMES:
Response Rate | Measured at week 16
Quality of life | Baseline to study completion
Progression free survival | Measured at week 16 and 52
Overall Survival | Measured at week 16 and 52

CONTACTS AND LOCATIONS:
Locations (10):
- United States (2):
  - Emory Clinic, Atlanta, Georgia
  - White Plains Hospital, White Plains, New York
- Israel (8):
  - Assaf Harofe Medical Center, Ẕerifin, Zerifin
  - HaEmek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv